CLINICAL TRIAL: NCT03988452
Title: Nucleosides And Darunavir/Dolutegravir In Africa (NADIA): a Randomised Controlled Trial of Darunavir Versus Dolutegravir and Tenofovir Versus Zidovudine in Second-line Antiretroviral Therapy Regimens for the Public Health Approach in Sub-Saharan Africa
Brief Title: Nucleosides And Darunavir/Dolutegravir In Africa
Acronym: NADIA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: JC3218
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir; dolutegravir; Zidovudine; Tenofovir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Darunavir/r Zidovudine Lamivudine (Active Comparator): Darunavir 800mg once daily Ritonavir 100mg once daily Zidovudine 300mg twice daily Lamivudine 150mg twice daily Combination given for 96 weeks
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Zidovudine; Drug: Lamivudine
- Darunavir/r Tenofovir Lamivudine (Experimental): Darunavir 800mg once daily Ritonavir 100mg once daily Tenofovir 300mg once daily Lamivudine 300mg once daily Combination given for 96 weeks
  Interventions: Drug: Darunavir; Drug: Ritonavir; Drug: Tenofovir; Drug: Lamivudine
- Dolutegravir Zidovudine Lamivudine (Experimental): Dolutegravir 50mg once daily Zidovudine 300mg twice daily Lamivudine 150mg twice daily Combination given for 96 weeks
  Interventions: Drug: Dolutegravir; Drug: Zidovudine; Drug: Lamivudine
- Dolutegravir Tenofovir Lamivudine (Experimental): Dolutegravir 50mg once daily Tenofovir 300mg once daily Lamivudine 300mg once daily Combination given for 96 weeks
  Interventions: Drug: Dolutegravir; Drug: Tenofovir; Drug: Lamivudine

INTERVENTIONS:
Drug: Darunavir — Antiretroviral therapy
  Arms: Darunavir/r Tenofovir Lamivudine; Darunavir/r Zidovudine Lamivudine
Drug: Ritonavir — Antiretroviral therapy
  Arms: Darunavir/r Tenofovir Lamivudine; Darunavir/r Zidovudine Lamivudine
Drug: Dolutegravir — Antiretroviral therapy
  Arms: Dolutegravir Tenofovir Lamivudine; Dolutegravir Zidovudine Lamivudine
Drug: Zidovudine — Antiretroviral therapy
  Arms: Darunavir/r Zidovudine Lamivudine; Dolutegravir Zidovudine Lamivudine
Drug: Tenofovir — Antiretroviral therapy
  Arms: Darunavir/r Tenofovir Lamivudine; Dolutegravir Tenofovir Lamivudine
Drug: Lamivudine — Antiretroviral therapy

SUMMARY:
This trial evaluates options for second-line antiretroviral therapy in patients failing on a non-nucleoside reverse transcriptase inhibitor (NNRTI) and tenofovir (TDF)-based first-line regimen in the setting of the public health approach in sub-Saharan Africa (with assumed substantial nucleoside reverse transcriptase inhibitor (NRTI) cross-resistance). The trial tests two hypotheses. Firstly that a regimen of dolutegravir (DTG) with two NRTIs is non-inferior to a regimen of ritonavir-boosted darunavir (DRV/r) with two NRTIs. Secondly that continuing an NRTI regimen of TDF and lamivudine (3TC) is non-inferior to switching to zidovudine (ZDV) and 3TC.

The trial is a parallel group, open-label, multi-centre, factorial (2X2) randomised, controlled trial. Patients will be randomised to either DTG or DRV/r with a second randomisation to ZDV and 3TC or TDF and 3TC. Treatment efficacy will be monitored by testing viral load (VL). Analyses will compare DRV/r with DTG; and ZDV/3TC with TDF/3TC by intention to treat analysis on the primary outcome parameter of plasma VL below 400 copies/ml at 48 weeks. Trial follow-up will continue to 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 12 years and above
2. Body weight at least 40kg
3. Taking a tenofovir plus lamivudine/emtricitabine plus NNRTI-based regimen continuously for a total period of at least 6 months
4. Good adherence to ART, defined as missing medication on no more than 3 days in the one month prior to screening. [Patients who do not have good adherence should be given adherence counselling and re-assessed after an interval of not less than 4 weeks].
5. HIV treatment failure defined by virological criteria (modified from WHO 2016 criteria); Viral load ≥ 1000 copies/ml at screening AND EITHER Viral load ≥ 1000 copies/ml on the previous test, taken after at least 6 months on ART, and at no more than 6 months prior to screening and at no less than 4 weeks prior to screening, with adherence counselling given after the previous test OR Viral load ≥ 1000 copies/ml on a confirmatory test taken no less than 4 weeks after screening with adherence counselling given after the screening test
6. If a woman of childbearing potential, must be willing to use effective contraception. [Childbearing potential is defined as being not premenarchal; not post-menopausal (> 12 months of spontaneous amenorrhea and ≥45 years of age); and not permanently sterilised].
7. Willing and able to provide written informed consent
8. Able to attend regular study follow-up visits

Exclusion Criteria:

1. Prior use of protease inhibitor or integrase inhibitor therapy
2. Requirement for concomitant medication with known major interactions with study drugs for which drug substitutions or dose alterations are not available or acceptable (if the patient requires rifamycin-based TB treatment, rifabutin must be available at the site).
3. Women who are currently pregnant or breastfeeding.
4. Severe hepatic impairment (with ascites and/or encephalopathy)
5. ALT > 5 times upper limit of normal
6. Estimated glomerular filtration rate (eGFR) < 50 ml/min/1.73m2 at screening calculated using the CKD-EPI equation
7. Current participation in another clinical trial or research protocol (may be permitted in some circumstances; but must first be discussed with the NADIA Chief Investigator)
8. Life expectancy of less than one month in the opinion of the treating physician

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Plasma viral load < 400 copies/ml at 48 weeks | 48 weeks

SECONDARY OUTCOMES:
Plasma viral load < 1000 copies/ml | 48 and 96 weeks
Plasma viral load < 400 copies/ml at 96 weeks | 96 weeks
Plasma viral load < 50 copies/ml | 48 and 96 weeks
Plasma viral load rebound (≥ 1000 copies/ml, confirmed) | 48 and 96 weeks
Plasma viral load rebound (≥ 400 copies/ml, confirmed) | 48 and 96 weeks
Plasma viral load rebound (≥ 50 copies/ml, confirmed) | 48 and 96 weeks
Viral load rebound (≥ 1000 copies/ml, confirmed) with ≥ 1 major resistance mutation (IAS list) to DRV or DTG | 48 and 96 weeks
Viral load rebound (≥ 1000 copies/ml, confirmed) with intermediate or high-level resistance (Stanford algorithm) to DRV or DTG | 48 and 96 weeks
Viral load rebound (≥ 1000 copies/ml, confirmed) with intermediate or high-level resistance (Stanford algorithm) to both zidovudine and tenofovir | 48 and 96 weeks
CD4+ cell count change from baseline | 48 and 96 weeks
Incident (new or recurrent) WHO stage 4 event | 48 and 96 weeks
Incident serious non-AIDS event | 48 and 96 weeks
Death | 48 and 96 weeks
Time to new or recurrent WHO Stage 4 event, serious non-AIDS event, or death | 96 weeks
Grade 3 or 4 clinical adverse events | 48 and 96 weeks
Grade 3 or 4 clinical adverse events (possibly, probably or definitely related to ART) | 48 and 96 weeks
Serious Adverse Events | 48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, MD, Study Director — National University of Singapore
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

REFERENCES:
- [Derived] Paton NI, Musaazi J, Kityo C, Walimbwa S, Hoppe A, Balyegisawa A, Asienzo J, Kaimal A, Mirembe G, Lugemwa A, Ategeka G, Borok M, Mugerwa H, Siika A, Odongpiny ELA, Castelnuovo B, Kiragga A, Kambugu A; NADIA Trial Team. Efficacy and safety of dolutegravir or darunavir in combination with lamivudine plus either zidovudine or tenofovir for second-line treatment of HIV infection (NADIA): week 96 results from a prospective, multicentre, open-label, factorial, randomised, non-inferiority trial. Lancet HIV. 2022 Jun;9(6):e381-e393. doi: 10.1016/S2352-3018(22)00092-3. Epub 2022 Apr 20. PMID 35460601
- [Derived] Paton NI, Musaazi J, Kityo C, Walimbwa S, Hoppe A, Balyegisawa A, Kaimal A, Mirembe G, Tukamushabe P, Ategeka G, Hakim J, Mugerwa H, Siika A, Asienzo J, Castelnuovo B, Kiragga A, Kambugu A; NADIA Trial Team. Dolutegravir or Darunavir in Combination with Zidovudine or Tenofovir to Treat HIV. N Engl J Med. 2021 Jul 22;385(4):330-341. doi: 10.1056/NEJMoa2101609. PMID 34289276